CLINICAL TRIAL: NCT00977886
Title: A Multiple Ascending Dose Study to Assess the Safety and Pharmacokinetics of Oral ELB353 in Healthy Male Volunteers - A Double-Blind, Randomized, Placebo-controlled, Sequential Group Study
Brief Title: Safety and Pharmacokinetics of ELB353 in Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biotie Therapies Corp. (Industry)
Responsible Party: CMO, Biotie Therapies Corp.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BTT70-CD018
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- ELB353 (Experimental)
  Interventions: Drug: ELB353

INTERVENTIONS:
Drug: Placebo — Oral, 10 days
  Arms: Placebo
Drug: ELB353 — Oral, 10 days
  Arms: ELB353

SUMMARY:
The purpose of this trial is to study the safety and tolerability of repeated oral doses of ELB353, to evaluate the plasma levels of ELB353 and to study their effect on substances mediating inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

* Concomitant medication
* Concomitant disease

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2009-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Adverse event frequency and intensity | 1 month

SECONDARY OUTCOMES:
Plasma levels of ELB353 | 1 month
Inflammatory transmitter response ex vivo | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Antero Kallio, MD, Study Director — Biotie Therapies Corp.
Locations (1):
- Biotie investigational site, Berlin, State of Berlin, Germany